CLINICAL TRIAL: NCT00060242
Title: Phase II Trial Of Combretastatin A-4 Phosphate (CA4P) In Advanced Anaplastic Carcinoma Of The Thyroid
Brief Title: Combretastatin A4 Phosphate in Treating Patients With Advanced Anaplastic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Panayiotis Savvides, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICC2302; P30CA043703 (NIH); CASE-CWRU-ICC-2302 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Head and Neck Cancer
Keywords: anaplastic thyroid cancer; recurrent thyroid cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms | interventions — fosbretabulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fosbretabulin disodium — Combretastatin A4 phosphate IV over 10 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 courses beyond documentation of the CR.
  Other Names: Combretastatin A4 phosphate

SUMMARY:
RATIONALE: Combretastatin A4 phosphate may stop the growth of anaplastic thyroid cancer by stopping blood flow to the tumor.

PURPOSE: This phase II trial is studying how well combretastatin A4 phosphate works in treating patients with advanced recurrent or metastatic anaplastic thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate of patients with advanced anaplastic thyroid cancer treated with combretastatin A4 phosphate.
* Determine whether this drug alters the natural history of anaplastic thyroid cancer, in terms of doubling the median survival from 4-6 months to 12 months, in these patients.
* Determine the safety profile of this drug in these patients.
* Correlate clinical response with pretreatment tumor microvessel density and immature vessel staining, changes in sICAM-1 levels over the course of treatment, and pharmacokinetic parameters in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive combretastatin A4 phosphate IV over 10 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 courses beyond documentation of the CR.

Patients are followed monthly.

PROJECTED ACCRUAL: A total of 32 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* anaplastic or poorly differentiated variant thyroid cancer, including 1 of the following:

  * Recurrent/regionally advanced disease no longer amenable to definitive curative surgery or radiotherapy
  * Untreated metastatic disease NOTE: *If original/diagnostic tumor blocks are unavailable, tumor must be accessible for pretreatment core needle biopsy
* Must have relapsed or progressed during or after prior combined modality therapy (e.g., systemic chemotherapy and radiotherapy) for regionally advanced (but not metastatic) disease
* Measurable or evaluable disease
* Patent trachea and airway by screening direct and indirect laryngoscopy* NOTE: *For patients with bulky thyroid/neck masses and/or suspected airway obstruction
* No active brain metastases, as evidenced by any of the following:

  * Symptomatic involvement
  * Cerebral edema by CT scan or MRI
  * Radiographic evidence of progression since definitive therapy
  * Continued requirement for corticosteroids

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin at least 8.5 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT and AST no greater than 3.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* LVEF at least 50% by MUGA
* EKG normal

  * No evidence of prior myocardial infarction (e.g., significant Q waves), QTc greater than 450 msec, or other clinically significant abnormalities
* No history of angina (even if controlled by medication)
* No congestive heart failure
* No uncontrolled atrial arrhythmias
* No clinically significant arrhythmias, including any of the following:

  * Conduction abnormalities
  * Nodal junctional arrhythmias and dysrhythmias
  * Sinus bradycardia or tachycardia
  * Supraventricular arrhythmias
  * Atrial fibrillation or flutter
  * Syncope or vasovagal episodes
* No significant heart wall abnormality or heart muscle damage by MUGA
* No uncontrolled hypertension (blood pressure consistently greater than 150 mm Hg systolic and 100 mm Hg diastolic regardless of medication)

  * Patients with previous hypertension are allowed provided there is clinical documentation of controlled blood pressure for 2 months prior to study enrollment
* No symptomatic peripheral vascular disease
* No symptomatic cerebrovascular disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No grade 2 or greater preexisting motor or sensory peripheral neuropathy
* No uncontrolled hypokalemia or hypomagnesemia
* No concurrent serious infection
* No other nonmalignant medical illness that is uncontrolled or whose control may be jeopardized by study therapy
* No psychiatric disorders or other conditions that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic therapy
* No concurrent immunotherapy
* No concurrent prophylactic colony-stimulating factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent hormonal therapy, except any of the following:

  * Gonadotropin-releasing hormone agonists for hormone-refractory prostate cancer
  * Hormone replacement therapy
  * Oral contraceptives
  * Megestrol for anorexia/cachexia

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy with progressive disease beyond radiation ports
* No prior radiotherapy to more than 30% of the bone marrow
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* More than 4 weeks since prior major surgery

Other

* At least 6 weeks since other prior therapy associated with delayed toxicity
* No prior therapy for metastatic disease
* No concurrent medication(s) known to prolong the QTc interval, unless medication(s) can be held for at least 72 hours before, during, and for at least 6 hours after study drug administration
* No other concurrent investigational therapy
* No other concurrent antineoplastic or cytotoxic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2003-02; Primary Completion 2007-02 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Median survival | every 8 weeks

SECONDARY OUTCOMES:
Objective disease response | every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Panayiotis Savvides, MD, Study Chair — Ireland Cancer Center at University Hosptials Case Medical Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Ireland Cancer Center at University Hosptials Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Mooney CJ, Nagaiah G, Fu P, Wasman JK, Cooney MM, Savvides PS, Bokar JA, Dowlati A, Wang D, Agarwala SS, Flick SM, Hartman PH, Ortiz JD, Lavertu PN, Remick SC. A phase II trial of fosbretabulin in advanced anaplastic thyroid carcinoma and correlation of baseline serum-soluble intracellular adhesion molecule-1 with outcome. Thyroid. 2009 Mar;19(3):233-40. doi: 10.1089/thy.2008.0321. PMID 19265494
- [Derived] Giri P, Batra PJ, Kumari A, Hura N, Adhikary R, Acharya A, Guchhait SK, Panda D. Development of QTMP: A promising anticancer agent through NP-Privileged Motif-Driven structural modulation. Bioorg Med Chem. 2023 Nov 15;95:117489. doi: 10.1016/j.bmc.2023.117489. Epub 2023 Oct 5. PMID 37816266